CLINICAL TRIAL: NCT05688228
Title: Description of the Evolution of Women's Sexuality After a Voluntary Interruption of Pregnancy
Brief Title: Voluntary Interruption of Pregnancy on Women's Sexuality
Acronym: VTOPSimpact
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/71
Record Dates: First submitted 2022-12-28; First posted 2023-01-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Abortion
Keywords: Abortion; Female sexuality; FSFI
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abortion: Adult women performing a medical or surgical abortion
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Female Sexual Function Index (FSFI) and self-administrative questionnaires on sexuality just after abortion and repeated at 1, 3 and 6 months

SUMMARY:
The impact on sexuality has been less studied and there is no French study on this subject and the rare studies are contradictory.

The aim of this study is to evaluate the impact of abortion (medical or surgical) on female sexuality, to look for a difference in the impact on sexuality according to the method used for the termination (medical or surgical) just after the procedure and at 1, 3 and 6 months and to look for risk factors and protective factors for the existence or occurrence of sexual dysfunction before and after abortion.

DETAILED DESCRIPTION:
The medical consequences of abortion are low. However, there is an undeniable emotional and psychological impact on these women (40-45% of anxiety-type symptoms, approximately 20% of depressive symptoms after the discovery of the pregnancy and 30% of emotional disorders, particularly anxiety, in the month following the abortion).

The impact on sexuality has been less studied and there is no French study on this subject and the rare studies are contradictory.

The aim of this study is to evaluate the impact of voluntary termination of pregnancy (medical or surgical) on female sexuality, to look for a difference in the impact on sexuality according to the method used for the termination (medical or surgical) just after the procedure and at 1, 3 and 6 months and to look for risk factors and protective factors for the existence or occurrence of sexual dysfunction before and after a termination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Patient performing a medical or surgical abortion
* Patient with health insurance
* No opposition to participation in the study

Exclusion Criteria:

* Patient who does not speak French and/or is illiterate
* Patient under legal protection
* Patient unable to complete the study procedures (no internet connection, no smart phone or tablet)
* Patient with diagnosed psychiatric comorbidities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women performing a medical or surgical abortion
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with sexual dysfunction | Month 6
  Sexual dysfunction is assessed using the Female Sexual Function Index (FSFI) questionnaire, which takes into account several aspects of female sexuality: desire, arousal, lubrication, orgasm, satisfaction and pain. The threshold for differentiating between patients with and without sexual dysfunction is 26.55

SECONDARY OUTCOMES:
Marital status | Baseline
  single, couple, married
Number of sexual partners in the last 12 months | Baseline
  Number of sexual partners via self-questionnaire : 1 ; from 2 to 5 ; from 6 to 10 ; from 11 to 15 ; from 16 to 20 ; up to 20
Number of sexual partners in the whole life | Baseline
  Number of sexual partners via self-questionnaire : 1 ; from 2 to 5 ; from 6 to 10 ; from 11 to 15 ; from 16 to 20 ; up to 20
Number of sexual partners in the last 4 weeks | Baseline
  Number of sexual partners via self-questionnaire : 0, 1, from 2 to 5, up to 5
Frequency of sexual activity in the last month before pregnancy discovery | Baseline, Month 1, Month 3, Month 6
  < 1 /month ; from 1 from 3 /month ; 1 /week ; twice /week ; 3 or more times /week
Existence of physical violence in the whole life | Baseline
  binary variable (yes/no)
Existence of psychological violence in the whole life | Baseline
  binary variable (yes/no)
Existence of sexual violence in the whole life | Baseline
  binary variable (yes/no)
Existence of psychological symptoms before pregnancy's discovery | Baseline
  asthenia, sadness, anxiety, guilt, none
Existence of psychological symptoms in the last month | Month 1, Month 3, Month 6
  asthenia, sadness, anxiety, guilt, none
Existence of sexual difficulties since pregnancy's discovery | Baseline
  Decreased desire, arousal, lubrication, quantity or quality of orgasms, sexual satisfaction or relationship with the partner, appearance or increase of pain during sexual intercourse, no change in these different areas of sexuality
Sexual activity the last month | Month 1, Month 3, Month 6
  Decreased sexual activity (fear of another pregnancy, waiting to start contraception, conflict with partner after abortion, other reason), Not concerned about decreased sexual activity
Contraception in the last month | Month 1, Month 3, Month 6
  none, removal/cycles, condoms, pill, intrauterine devic, implant, ring/patch, other

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No